CLINICAL TRIAL: NCT00428948
Title: A Phase 3, Multi-center, Double-blind, Placebo-controlled, Parallel-arm Trial to Determine Long-term Safety and Efficacy of Oral Tolvaptan Tablets Regimens in Adult Subjects With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Tolvaptan Phase 3 Efficacy and Safety Study in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Acronym: TEMPO3:4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-04-251; 2006-002768-24 (EudraCT Number)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Kidney Disease, Autosomal Dominant
Keywords: ADPKD; Polycystic; kidney; ADPKD (Autosomal Dominant Polycystic Kidney Disease)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan (Experimental): Participants received the highest tolerated split-dose regimen (upon awakening and 9 hours later) of tolvaptan 45/15 mg, 60/30 mg, or 90/30 mg orally for 36 months.
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Participants received placebo (upon awakening and 9 hours later) orally for 36 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan was supplied as tablets.
  Other Names: OPC-41061; OPC-156
  Arms: Tolvaptan
Drug: Placebo — Placebo was supplied as tablets.
  Arms: Placebo

SUMMARY:
This study's purpose is to evaluate the long-term safety and efficacy of tolvaptan versus placebo in patients with ADPKD.

DETAILED DESCRIPTION:
This study evaluated whether or not tolvaptan is potentially beneficial, while maintaining an adequate safety profile, by reducing the rate of total kidney volume increase, while impacting the onset, severity, and progression of other important consequences of ADPKD.

During the 3-week titration phase, tolvaptan or placebo was titrated in weekly intervals from lowest to highest tolerated levels given in split-dose regimens of 45/15 mg, 60/30 mg and 90/30 mg orally upon awakening and approximately 9 hours later. As soon as a subject could not tolerate a given dose, the titration phase was over and the maintenance phase began at the dose level tolerated. The maintenance phase lasted to Month 36. Subjects were able to titrate down at any point during the study. Subjects were able to titrate up during the maintenance phase with Medical Monitor approval.

ELIGIBILITY:
Inclusion Criteria:

* Legal adult age and able to give Informed Consent.
* Adult subjects with a diagnosis of ADPKD. A diagnosis of ADPKD (age 18 or 20-50) required several cysts in each kidney (3 if by sonography, 5 if by CT or MRI) in those with a family history of ADPKD and 10 cysts (by any radiologic method) in each kidney and exclusion of other cystic kidney diseases if there was no family history.
* Willingness to comply with reproductive precautions, if female.
* Estimated creatinine clearance ≥ 60 mL/min. Estimated from serum creatinine during screening using Cockcroft-Gault with correction for gender and race, where possible.
* Rapidly progressive kidney growth (total volume ≥ 750 cc) by magnetic resonance imaging (MRI) at randomization.

Exclusion Criteria:

* Prior exposure to tolvaptan or other experimental PKD therapies.
* Currently taking medication for purpose of affecting PKD cysts.
* Women who are breast feeding and females of childbearing potential who are not using acceptable contraceptive methods.
* In the opinion of the study investigator or sponsor may present a safety risk or confound study objectives.
* Patients who are unlikely to adequately comply with study procedures.
* Patients having contraindications to MRI.
* Patients taking medications or having any illnesses likely to affect ADPKD outcomes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1445 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Torres, MD, PhD, Principal Investigator — Mayo Medical Center; Frank Czerwiec, MD, PhD, Study Director — Otsuka Pharmaceutical Development and Commercialization, Inc.; Osamu Sato, Study Director — Otsuka Pharmaceutical Corporation, Ltd. Japan
Locations (133):
- United States (30):
  - Coastal Clinical Research, Mobile, Alabama
  - University of South Alabama, Mobile, Alabama
  - Apex Research of Riverside, Riverside, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Coastal Nephrology Associates Research Center, LLC, Port Charlotte, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Renal Associates of Baton Rough, L.L.C., Baton Rouge, Louisiana
  - John Hopkins School of Medicine, Baltimore, Maryland
  - Tufts- New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Medical Center, Rochester, Minnesota
  - Erie County Medical Center, Buffalo, New York
  - Nephrology Associates of Westchester, Hawthorne, New York
  - The Rogosin Institute, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, UNC, Kidney Center, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Kidney and Hypertension Center, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case, Cleveland, Ohio
  - Northwest Renal Clinic, Inc., Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Charleston Nephrology Associates, Charleston, South Carolina
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Nephrology Clinical Research Center, Charlottesville, Virginia
- Argentina (5):
  - Instituto de Nefrología, Nefrology SA, Buenos Aires
  - Hospital Municipal de Vicente Lopez, Dr Bernardo Houssay, Buenos Aires
  - Hosptial Universitario Austral, Buenos Aires
  - Sanatorio Allende, Córdoba
  - Hospital Privado-Centro Medico de Cordoba, Córdoba
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - Queen Elizebeth Hospital, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - Royal Melbourne Hospital, Melbourne
  - Melbourne Renal Research Group, Melbourne
  - Royal Perth Hospital, Perth
  - Royal North Shore Hospital, Sydney
  - Westmead Hospital, Sydney
- Belgium (3):
  - UZ Brussel, Brussels
  - Ucl-St Luc, Brussels
  - UZ Gent, Ghent
- Canada (3):
  - Queen Elizabeth II Health Science Center, Division of Nephrology, Halifax, Nova Scotia
  - Royal Victoria Hospital, Montreal, Quebec
  - Hospital du Sacre- Coeur de Montreal, Montreal, Quebec
- Denmark (2):
  - Herlev Amtssygehus, Herlev
  - Odense Universitetshospital, Odense
- France (9):
  - CHU-Hopital Pellegrin, Bordeaux
  - CHU - Hôpital Clémenceau, Caen
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Conception, Marseille
  - CHU - Hôpital Lapeyronie, Montpellier
  - Hopital Bichat-Claude Bernard, Paris
  - Centre Hospitalier Universitaire, Reims
  - CHU - Hôpital Nord, Saint-Etienne
  - Hopital Rangueil, Toulouse
- Germany (6):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Nephrologische Gemeinschaftspraxis/Dialysezentrum, Düsseldorf
  - Klinik für Nieren- und Hochdruckkrankheiten, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätskliniken Heidelberg, Heidelberg
  - UH Erlangen/Nürnberg, Nuremberg
- Italy (5):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Università Vita e Salute, Ospedale San Raffaele, Milan
  - Policlinico di Modena, Modena
  - Policlinico, Napoli
  - IRCCS Fondazione Salvatore Maugeri, Pavia
- Japan (30):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tokai University Hospital, Isehara, Kanagawa
  - Toranomon Hospital Kajigaya, Kawasaki, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Shuwa General Hospital, Kasukabe, Saitama
  - Saitama Medical Center, Kawagoe, Saitama
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Jichi Medical School Hospital, Shimotsuke, Tochigi
  - Tokyo Medical & Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Kyusyu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima University Hospital, Hiroshima
  - Kumamoto Univeristy Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Ohno Memorial Hospital, Osaka
  - Saitama Medical Center Jichi Medical University, Saitama
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - UMCG Groningen, Groningen
- Poland (11):
  - Oddział Nefrologiczny Stacja Dializ, Ciechanów
  - Akademickie Centrum Kliniczne AMG, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Akademickie Centrum Kliniczne AMG, Gdansk
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Szpital Uniwersytecki w Krakowie, Krakow
  - SOP ZOZ Uniwersytecki Szpital Kliniczny, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Klinika Chorób Wewnętrznych i Nefrologii, Warsaw
  - Szpital Praski p.w. Przemienienia Panskiego, Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Warsaw
  - Szpital Praski, Samodzielny Publiczny ZOZ, Warsaw
  - Międzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - Akademicki Szpital Kliniczny im J Mikulicza Radeckiego, Wroclaw
- Romania (3):
  - Spitalul Clinic de Nefrologie Dr. Carol Davila, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic "C.I.Parhon", Iași
- Russia (5):
  - Kemerovo Medical Academy, Regional Clinical Hospital, Kemerovo
  - City Clinical Hospital #52, Moscow
  - City Mariinskiy Hospital, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Tomsk Regional Clinical Hospital, Tomsk
- United Kingdom (11):
  - Belfast City Hospital, Belfast
  - Oueen Elizabeth Hospital, Birmingham
  - Sussex Renal Unit Royal Sussex County Hospital, Brighton
  - Uhcw Mhs Trust, Coventry
  - Royal Infirmary, Edinburgh
  - Raigmore Hospital, Inverness
  - Royal Free and University College Medical School, London
  - King's College Hospital, London
  - St. George's Hospital, London
  - Royal Hallamshire Hospital, Sheffield
  - Morriston Hospital, Swansea

REFERENCES:
- [Background] Gattone VH 2nd, Wang X, Harris PC, Torres VE. Inhibition of renal cystic disease development and progression by a vasopressin V2 receptor antagonist. Nat Med. 2003 Oct;9(10):1323-6. doi: 10.1038/nm935. Epub 2003 Sep 21. PMID 14502283
- [Background] Torres VE, Wang X, Qian Q, Somlo S, Harris PC, Gattone VH 2nd. Effective treatment of an orthologous model of autosomal dominant polycystic kidney disease. Nat Med. 2004 Apr;10(4):363-4. doi: 10.1038/nm1004. Epub 2004 Feb 29. PMID 14991049
- [Background] Torres VE, Meijer E, Bae KT, Chapman AB, Devuyst O, Gansevoort RT, Grantham JJ, Higashihara E, Perrone RD, Krasa HB, Ouyang JJ, Czerwiec FS. Rationale and design of the TEMPO (Tolvaptan Efficacy and Safety in Management of Autosomal Dominant Polycystic Kidney Disease and its Outcomes) 3-4 Study. Am J Kidney Dis. 2011 May;57(5):692-9. doi: 10.1053/j.ajkd.2010.11.029. Epub 2011 Feb 17. PMID 21333426
- [Background] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Grantham JJ, Higashihara E, Perrone RD, Krasa HB, Ouyang J, Czerwiec FS; TEMPO 3:4 Trial Investigators. Tolvaptan in patients with autosomal dominant polycystic kidney disease. N Engl J Med. 2012 Dec 20;367(25):2407-18. doi: 10.1056/NEJMoa1205511. Epub 2012 Nov 3. PMID 23121377
- [Background] Watkins PB, Lewis JH, Kaplowitz N, Alpers DH, Blais JD, Smotzer DM, Krasa H, Ouyang J, Torres VE, Czerwiec FS, Zimmer CA. Clinical Pattern of Tolvaptan-Associated Liver Injury in Subjects with Autosomal Dominant Polycystic Kidney Disease: Analysis of Clinical Trials Database. Drug Saf. 2015 Nov;38(11):1103-13. doi: 10.1007/s40264-015-0327-3. PMID 26188764
- [Background] Kher A. Tolvaptan in autosomal dominant polycystic kidney disease. N Engl J Med. 2013 Mar 28;368(13):1257-8. doi: 10.1056/NEJMc1300762. No abstract available. PMID 23534570
- [Background] Spital A. Tolvaptan in autosomal dominant polycystic kidney disease. N Engl J Med. 2013 Mar 28;368(13):1257. doi: 10.1056/NEJMc1300762. No abstract available. PMID 23534569
- [Background] Torres VE, Gansevoort RT, Czerwiec FS. Tolvaptan in autosomal dominant polycystic kidney disease. N Engl J Med. 2013 Mar 28;368(13):1259. doi: 10.1056/NEJMc1300762. No abstract available. PMID 23534568
- [Background] Jouret F, Krzesinski JM. Tolvaptan in autosomal dominant polycystic kidney disease. N Engl J Med. 2013 Mar 28;368(13):1258-9. doi: 10.1056/NEJMc1300762. No abstract available. PMID 23534572
- [Background] Sexton DJ. Tolvaptan in autosomal dominant polycystic kidney disease. N Engl J Med. 2013 Mar 28;368(13):1258. doi: 10.1056/NEJMc1300762. No abstract available. PMID 23534571
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Ivaturi V, Gobburu J, Leslie B, Wang X, Jadhav P. Urine Osmolality Is a Potential Marker of Longer-Term Efficacy of Tolvaptan in Autosomal Dominant Polycystic Kidney Disease: A Post Hoc Analysis. Kidney360. 2024 Jul 1;5(7):996-1001. doi: 10.34067/KID.0000000000000485. Epub 2024 Jun 10. PMID 38857379
- [Derived] Mochizuki T, Matsukawa M, Tanaka T, Jiang H. Initial eGFR Changes Predict Response to Tolvaptan in ADPKD. Kidney360. 2024 Apr 1;5(4):522-528. doi: 10.34067/KID.0000000000000404. Epub 2024 Feb 28. PMID 38414126
- [Derived] Gobburu J, Ivaturi V, Wang X, Shoaf SE, Jadhav P, Perrone RD. Comparing Effects of Tolvaptan and Instruction to Increase Water Consumption in ADPKD: Post Hoc Analysis of TEMPO 3:4. Kidney360. 2023 Dec 1;4(12):1702-1707. doi: 10.34067/KID.0000000000000302. Epub 2023 Nov 21. PMID 37986188
- [Derived] Lioudis M, Zhou X, Davenport E, Nunna S, Krasa HB, Oberdhan D, Fernandes AW. Effects of tolvaptan discontinuation in patients with autosomal dominant polycystic kidney disease: a post hoc pooled analysis. BMC Nephrol. 2023 Jun 22;24(1):182. doi: 10.1186/s12882-023-03247-6. PMID 37349694
- [Derived] Alpers DH, Lewis JH, Hunt CM, Freston JW, Torres VE, Li H, Wang W, Hoke ME, Roth SE, Westcott-Baker L, Estilo A. Clinical Pattern of Tolvaptan-Associated Liver Injury in Trial Participants With Autosomal Dominant Polycystic Kidney Disease (ADPKD): An Analysis of Pivotal Clinical Trials. Am J Kidney Dis. 2023 Mar;81(3):281-293.e1. doi: 10.1053/j.ajkd.2022.08.012. Epub 2022 Sep 30. PMID 36191725
- [Derived] Nowak KL, Steele C, Gitomer B, Wang W, Ouyang J, Chonchol MB. Overweight and Obesity and Progression of ADPKD. Clin J Am Soc Nephrol. 2021 Jun;16(6):908-915. doi: 10.2215/CJN.16871020. Epub 2021 Jun 11. PMID 34117082
- [Derived] Heida JE, Gansevoort RT, Torres VE, Devuyst O, Perrone RD, Lee J, Li H, Ouyang J, Chapman AB. The Effect of Tolvaptan on BP in Polycystic Kidney Disease: A Post Hoc Analysis of the TEMPO 3:4 Trial. J Am Soc Nephrol. 2021 Jul;32(7):1801-1812. doi: 10.1681/ASN.2020101512. Epub 2021 Apr 22. PMID 33888577
- [Derived] Bennett H, McEwan P, Hamilton K, O'Reilly K. Modelling the long-term benefits of tolvaptan therapy on renal function decline in autosomal dominant polycystic kidney disease: an exploratory analysis using the ADPKD outcomes model. BMC Nephrol. 2019 Apr 23;20(1):136. doi: 10.1186/s12882-019-1290-5. PMID 31014270
- [Derived] McEwan P, Bennett Wilton H, Ong ACM, Orskov B, Sandford R, Scolari F, Cabrera MV, Walz G, O'Reilly K, Robinson P. A model to predict disease progression in patients with autosomal dominant polycystic kidney disease (ADPKD): the ADPKD Outcomes Model. BMC Nephrol. 2018 Feb 13;19(1):37. doi: 10.1186/s12882-017-0804-2. PMID 29439650
- [Derived] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Perrone RD, Dandurand A, Ouyang J, Czerwiec FS, Blais JD; TEMPO 4:4 Trial Investigators. Multicenter, open-label, extension trial to evaluate the long-term efficacy and safety of early versus delayed treatment with tolvaptan in autosomal dominant polycystic kidney disease: the TEMPO 4:4 Trial. Nephrol Dial Transplant. 2018 Mar 1;33(3):477-489. doi: 10.1093/ndt/gfx043. PMID 28379536
- [Derived] Muto S, Kawano H, Higashihara E, Narita I, Ubara Y, Matsuzaki T, Ouyang J, Torres VE, Horie S. The effect of tolvaptan on autosomal dominant polycystic kidney disease patients: a subgroup analysis of the Japanese patient subset from TEMPO 3:4 trial. Clin Exp Nephrol. 2015 Oct;19(5):867-77. doi: 10.1007/s10157-015-1086-2. Epub 2015 Feb 7. PMID 25663351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat population: All randomized participants.
Period: Overall Study
Arm/Group | Tolvaptan | Placebo
Started | 961 | 484
Received Treatment | 961 | 483
Completed | 740 | 417
Not Completed | 221 | 67
Not completed — Lost to Follow-up | 15 | 8
Not completed — Adverse Event | 148 | 24
Not completed — Subject Met Withdrawal Criteria | 4 | 0
Not completed — Investigator Withdrew Subject | 3 | 4
Not completed — Subject Withdrew Consent | 50 | 30
Not completed — Protocol Deviation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan | Placebo | Total
Number analyzed (Participants) | 961 | 484 | 1445
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (7.1) | 38.8 (7.1) | 38.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 466 | 233 | 699
  Male | 495 | 251 | 746

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change Per Year in Total Kidney Volume From Baseline to Month 36
Description: Kidney volume was assessed in T1-weighted magnetic resonance images collected at each study site and sent to a central reviewing facility. At the central reviewing facility, blinded radiologists used proprietary software to measure the volume of both kidneys.
Time Frame: Baseline to Month 36
Population: Intent-to-treat population: All randomized participants who had Baseline and post-baseline observations of total kidney volume. Only participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change per year
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 819 | 458
Percentage change per year | 2.777 (5.659) | 5.608 (5.330)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in the percentage change per year in total kidney volume between the tolvaptan group and the placebo group; Test type: Superiority or Other; p < 0.0001, Linear mixed model; Mean Difference (Final Values) = -2.708, 95% CI 2-sided [-3.269 to -2.147] — The variance of the random effect intercept was zero and resulted in a non-positive, definite variance-covariance matrix for the random effects

2. Secondary Outcome: Number of ADPKD Clinical Progression Events Per 100 Follow-up Years From Baseline to Month 36
Description: These ADPKD events in the key secondary Outcome Measure were selected on the basis of their potential relationship to progressing cystogenesis. Reducing the rate of cyst development and expansion would likely slow the progression of ADPKD. The 4 events were: (1) Onset or progression of hypertension (someone is hypertensive if they have > 139 mmHg systolic blood pressure [BP], > 89 mmHg diastolic BP, or if they are taking antihypertensive medication at any BP level); (2) severe renal pain requiring medical intervention; (3) worsening albuminuria (by category, see below); and (4) worsening renal function, defined as a 25% decrease in 1/serum creatinine from Baseline. Albuminuria was assessed using spot urine albumin/creatinine ratio measurements (all measurements in mg/mmol). Categories included normal (< 2.8 female or < 2.0 male), microalbuminuria (2.8-28 female or 2.0-20 male), and overt proteinuria (> 28 female or > 20 male.
Time Frame: Baseline to Month 36
Population: Intent-to-treat population: All randomized participants. Only participants with available data were included in the analysis.
Measure: Number; unit: Events/100 follow-up years
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 961 | 483
Events/100 follow-up years | 43.94 | 50.04
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in the ADPKD clinical progression events/100 follow-up years between the tolvaptan group and the placebo group; Test type: Superiority or Other; p = 0.0095, Recurrent event analysis; Hazard Ratio (HR) = 0.865, 95% CI 2-sided [0.775 to 0.965] — Tolvaptan divided by placebo

3. Secondary Outcome: Change in Renal Function Per Year From Week 3 to Month 36
Description: Renal function was assessed using serum creatinine measurements and was estimated using 1/serum creatinine. The formula for 1/serum creatinine is: 1/Pcr, where Pcr = serum creatinine concentration (mg/dL). The change in renal function per year was based on the slope of change, obtained by regressing renal function data against time by subject.
Time Frame: Week 3 to Month 36
Population: Intent-to-treat population: All randomized participants with at least 4 months of follow-up. Only participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: (mg/mL)^-1 per year
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 842 | 464
(mg/mL)^-1 per year | -2.555 (9.767) | -3.682 (6.361)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in the change in renal function per year between the tolvaptan group and the placebo group; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Derived from testing the time treatment interaction using linear mixed model in which both intercept and slope are fixed and random effects; Difference in slope = 0.977, 95% CI 2-sided [0.597 to 1.357]

4. Secondary Outcome: Change in Mean Arterial Blood Pressure Per Year in Non-hypertensive Participants From Baseline to Month 36
Description: For participants who were non-hypertensive (systolic BP ≤ 139 mmHg and diastolic BP ≤ 89 mmHg without taking antihypertensive medications) at baseline, mean arterial blood pressure was measured at scheduled clinic visits up to the point of exposure to antihypertensive therapy for any reason. The change in mean arterial blood pressure per year was based on the slope of blood pressure, obtained by regressing blood pressure against time by subject.
Time Frame: Baseline to Month 36
Population: Intent-to-treat population: All randomized participants with at least 4 months of follow-up. Only non-hypertensive participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 74
mmHg | 2.561 (9.798) | 2.592 (7.095)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in mean arterial blood pressure in non-hypertensive participants between the tolvaptan group and the placebo group; Test type: Superiority or Other; p = 0.5520, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Difference in slope = -0.246, 95% CI 2-sided [-1.059 to 0.566] — Placebo minus tolvaptan

5. Secondary Outcome: Area Under the Concentration-time Curve of Change in Renal Pain From Baseline to Month 36
Description: Change from baseline in renal pain was assessed by a 0 to 10 pain scale as average area under the concentration-time curve (AUC) between baseline and the last trial visit or the last visit prior to initiating medical (eg, narcotic or anti-nociceptives [eg, tricyclic antidepressants]) or surgical therapy for pain. In the pain scale, score 0 represented no pain at all and score 10 represented the worst pain. A negative change score indicates less pain. AUC of renal pain was derived from renal pain scores within treatment period and was calculated using the trapezoidal rule, by dividing the number of days between the first and last assessment.
Time Frame: At screening, Baseline, Day 1, every 4 months up to month 36/early tremination (ET), follow-up visit 1 and 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 926 | 467
units on a scale | -0.00 (1.29) | 0.08 (1.43)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in the change in renal pain between the tolvaptan group and the placebo group; Test type: Superiority or Other; p = 0.1604, ANCOVA; The analysis included baseline renal pain as a covariate; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.20 to 0.03] — Derived from ANCOVA with factors of treatment and baseline stratification factor interaction and covariate renal pain baseline

6. Secondary Outcome: Number of Hypertensive Events Per 100 Follow-up Years in Non-hypertensive Participants From Baseline to Month 36
Description: A hypertensive event was defined as a change from non-hypertensive (systolic BP ≤ 139 mmHg and diastolic BP ≤ 89 mmHg without taking antihypertensive medications) status to 1 of 3 conditions: (1) High pre-hypertensive (systolic BP [sBP] > 129 mmHg and/or diastolic BP [dBP] > 84 mmHg), (2) hypertensive (sBP > 139 mmHg and/or dBP > 89 mmHg), or (3) requiring antihypertensive therapy.
Time Frame: Baseline to Month 36
Population: as for outcome 4
Measure: Number; unit: Events/100 follow-up years
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 174 | 79
Events/100 follow-up years | 31.80 | 29.60
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in the hypertensive events per 100 follow-up years in non-hypertensive participants between the tolvaptan group and the placebo group; Test type: Superiority or Other; p = 0.9704, Recurrent event analysis; Hazard Ratio (HR) = 0.996, 95% CI 2-sided [0.805 to 1.233] — Derived from rate and mean model of time to recurrent event analysis with factor treatment

7. Secondary Outcome: Percentage of Participants With a Clinically Sustained Decrease of Blood Pressure Leading to a Sustained Reduction in Antihypertensive Therapy From Baseline to Month 36
Time Frame: Baseline to Month 36
Population: Intent-to-treat population: All randomized participants with at least 4 months of follow-up. Only participants taking antihypertensive medication at Baseline with available data were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 481 | 267
Percentage of participants | 6.24 | 5.62
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; The null hypothesis was that there was no difference in the percentage of participants with a clinically sustained decrease of blood pressure leading to a sustained reduction in antihypertensive therapy between the tolvaptan group and the placebo group; Test type: Superiority or Other; p = 0.7532, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.100, 95% CI 2-sided [0.602 to 2.017] — Tolvaptan divided by placebo

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent, throughout the 3 year treatment period and up to 42 days after the last dose of study medication
Description: Safety population: All randomized participants who received study treatment. One participant in the placebo group did not receive study treatment and was not included in the safety population.
Arm/Group | Tolvaptan | Placebo
Serious Adverse Events (participants affected / at risk) | 177/961 | 95/483
Other Adverse Events (participants affected / at risk) | 793/961 | 372/483
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=961) | Placebo (N=483)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Multiple endocrine adenomatosis (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 0
Uveitis (Eye disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 8 | 2
Exercise tolerance decreased (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Pyrexia (General disorders) | 0 | 2
Thirst (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Hepatic pain (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 4
Arthritis bacterial (Infections and infestations) | 1 | 1
Bartholin's abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatic cyst infection (Infections and infestations) | 0 | 2
Hepatitis B (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 2 | 0
Liver abscess (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Mycoplasma infection (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Pyelonephritis (Infections and infestations) | 5 | 5
Renal cyst infection (Infections and infestations) | 6 | 4
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Syphilis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3
Urogenital infection bacterial (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Induced abortion haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 9 | 2
Aspartate aminotransferase increased (Investigations) | 9 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 2 | 1
Transaminases increased (Investigations) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Ligament pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 0
Intracranial aneurysm (Nervous system disorders) | 3 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 0
Migraine with aura (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Vertebral artery dissection (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 2
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 3 | 4
Renal cyst ruptured (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 4
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Asthenospermia (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Hysterocele (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 3 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0
Ovarian torsion (Reproductive system and breast disorders) | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 3 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 3 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=961) | Placebo (N=483)
Anaemia (Blood and lymphatic system disorders) | 30 | 26
Abdominal distension (Gastrointestinal disorders) | 49 | 17
Abdominal pain (Gastrointestinal disorders) | 63 | 32
Abdominal pain upper (Gastrointestinal disorders) | 63 | 43
Constipation (Gastrointestinal disorders) | 81 | 12
Diarrhoea (Gastrointestinal disorders) | 133 | 54
Dry mouth (Gastrointestinal disorders) | 154 | 60
Dyspepsia (Gastrointestinal disorders) | 78 | 16
Nausea (Gastrointestinal disorders) | 101 | 59
Vomiting (Gastrointestinal disorders) | 81 | 40
Asthenia (General disorders) | 58 | 27
Fatigue (General disorders) | 132 | 47
Oedema peripheral (General disorders) | 88 | 46
Pyrexia (General disorders) | 45 | 41
Thirst (General disorders) | 532 | 99
Bronchitis (Infections and infestations) | 59 | 36
Gastroenteritis (Infections and infestations) | 55 | 22
Influenza (Infections and infestations) | 78 | 38
Nasopharyngitis (Infections and infestations) | 221 | 111
Sinusitis (Infections and infestations) | 56 | 23
Upper respiratory tract infection (Infections and infestations) | 87 | 42
Urinary tract infection (Infections and infestations) | 87 | 65
Blood creatinine increased (Investigations) | 140 | 71
Decreased appetite (Metabolism and nutrition disorders) | 69 | 5
Polydipsia (Metabolism and nutrition disorders) | 100 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 138 | 90
Myalgia (Musculoskeletal and connective tissue disorders) | 52 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 27
Dizziness (Nervous system disorders) | 108 | 42
Headache (Nervous system disorders) | 243 | 123
Insomnia (Psychiatric disorders) | 55 | 23
Haematuria (Renal and urinary disorders) | 71 | 68
Nocturia (Renal and urinary disorders) | 281 | 63
Pollakiuria (Renal and urinary disorders) | 222 | 26
Renal pain (Renal and urinary disorders) | 266 | 172
Cough (Respiratory, thoracic and mediastinal disorders) | 78 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 50 | 18
Dry skin (Skin and subcutaneous tissue disorders) | 49 | 9
Hypertension (Vascular disorders) | 324 | 178
Polyuria (Renal and urinary disorders) | 369 | 83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No